CLINICAL TRIAL: NCT05729958
Title: Total Ankle Replacement Using Guides, Expert Versus Trainee
Acronym: TARGET
Status: Not yet recruiting | Type: Observational
Sponsor: Centre for Orthopaedic Research Alkmaar (Other)
Collaborators: Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, Joyce L Benner, PhD, Principal Investigator, Centre for Orthopaedic Research Alkmaar
Other Study IDs: NL83260.018.22
Record Dates: First submitted 2023-01-17; First posted 2023-02-15 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Ankle Osteoarthritis
Keywords: Arthroplasty; Patient-specific Instrumentation
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT scan — CT scan of the involved ankle

SUMMARY:
Patient Specific Instrumentation (PSI) is thought to quicken joint arthroplasty surgery by shortening the operation time and improving alignment. Studies about the learning curve of PSI for total ankle replacement (TAR) are lacking because it was only introduced in 2014.

The investigators believe that PSI could give a beginning ankle surgeon, or surgeons new to TAR, an advantage since PSI facilitates the complex TAR procedure. As such, the availability of TAR in Dutch patients with end-stage ankle osteoarthritis could be extended. To estimate this potential of PSI for TAR, the investigators aim (1) to compare the alignment accuracy of TAR performed using PSI between a beginning and an experienced orthopedic surgeon, and (2) to determine the learning curve of TAR performed using PSI for a beginning foot and ankle specialist by comparing the operative time, complications, and patient-reported outcomes with those of an experienced specialist.

DETAILED DESCRIPTION:
Total ankle replacement (TAR) as treatment of end-stage osteoarthritis of the ankle is gaining popularity past few years, resulting in a growing number of TAR placed each year. This is an important progression because osteoarthritis of the ankle is suggested to be as disabling as chronic kidney injury or heart failure. Though TAR is proposed to be superior to ankle arthrodesis (AA) with regard to patient quality of life, it is not commonly available in the Netherlands. Merely 149 TARs were registered nationally in 2020.

Patient Specific Instrumentation (PSI) is thought to quicken the process by shortening the operation time and improving alignment. Though the literature is submerged in studies about the learning curves of PSI and TAR, research about the learning curve of PSI TAR is lacking because it was only introduced in 2014. Preliminary results showed that the use of PSI resulted in lower average pain scores and earlier recovery compared to TAR using standard instrumentation. Yet the absolute advantage of PSI was not established because of limited research. Furthermore, all previous studies were performed by skilled surgeons to eliminate the bias of inexperience.

The investigators believe that PSI could give a beginning ankle surgeon, or surgeon new to TAR, an advantage since PSI facilitates the complex TAR procedure. As such, the availability of TAR in Dutch patients with end-stage ankle osteoarthritis could be extended. To estimate this potential of PSI for TAR, the investigators aim (1) to compare the alignment accuracy of TAR performed using PSI between a beginning and an experienced orthopedic surgeon, and (2) to determine the learning curve of TAR performed using PSI for a beginning foot and ankle specialist by comparing the operative time, complications, and patient-reported outcomes with those of an experienced specialist. It is hypothesized that the alignment of PSI TAR performed by a beginning orthopedic surgeon does not significantly differ from one performed by an experienced surgeon. Furthermore, it is hypothesized that the operative time, complications, and patient-reported outcomes do not significantly differ between a beginning and an experienced orthopedic surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patient can understand the study's meaning and is willing to sign the study-specific Informed Patient Consent Form.
* Patient received the implantation of Infinity or Inbone prosthesis using PROPHECY PSI for primary TAR in 2022.
* There are at least 3 months of follow-up data for this patient.
* Patient can lay still during the length of duration of the CT-scan.

Exclusion Criteria:

* If per-operative the use of the PSI guides was abandoned.
* Patients that underwent revision surgery (defined as original tibia of talar component change or removal).
* Patients that endured other diseases that significantly impacted the post-operative period following TAR (e.g. amputation, severe extremity dysfunction due to a neurological or vascular impairment or trauma).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that received primary TAR pre-operatively planned using PROPHECY PSI in 2022. Both traumatic and non-traumatic osteoarthritis are included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative TAR component accuracy | 2-year follow-up assessment
  Difference between the planned and obtained (anterior and sagittal) tibia angles.

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score (FAOS) | 2-year follow-up assessment
  The FAOS was developed to assess the patients' opinion about a variety of foot and ankle-related problems. FAOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport(Rec), and foot and ankle-related Quality of Life (QOL). The last week is taken into consideration when answering the questionnaire. Standardized answer options are given (% Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Foot Function Index (FFI) | 2-year follow-up assessment
  The FFI (questionnaire) consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability, and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), which best describes their foot over the past week.
  The pain subcategory consists of 9 items and measures foot pain in different situations, such as walking barefoot versus walking with shoes.
  The disability subcategory consists of 9 items and measures difficulty performing various functional activities because of foot problems, such as difficulty climbing stairs.
  The activity limitation subcategory consists of 5 items and measures limitations in activities because of foot problems, such as staying in bed all day. Recorded on a visual analog scale (VAS), scores range from 0 to 100 mm, with higher scores indicating worse pain.
American Orthopedic Foot and Ankle Score (AOFAS) | 2-year follow-up assessment
  This clinical rating system combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient (to assess sagittal motion, hindfoot motion, ankle-hindfoot stability, and alignment of the ankle-hindfoot). The scale includes 9 items that can be divided into 3 subscales (pain, function, and alignment). Pain consists of 1 item with a maximal score of 40 points, indicating no pain. Function consists of 7 items with a maximal score of 50 points, indicating full function. Alignment consists of 1 item with a maximal score of 10 points, indicating good alignment. The maximal score is 100 points, indicating no symptoms or impairments.

OTHER OUTCOMES:
Complications | 2-year follow-up
  Complications following TAR, and any reoperation or revision surgery

IPD SHARING:
Plan to Share IPD: Undecided